CLINICAL TRIAL: NCT05481138
Title: Wearable Augmented Prediction of Burnout in Nurses: A Synergy of Engineering, Bioethics, Nursing and Wellness Sciences
Brief Title: Predicting Burnout in Nurses
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Arjun P. Athreya, Principal Investigator, Mayo Clinic
Other Study IDs: 22-000447; R01NR020362-01 (NIH)
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Burnout, Healthcare Workers
Keywords: Registered Nurses; Artificial intelligence; Wearable
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to develop a technology to predict burnout in RNs by measuring workplace, psychological, and physiological factors experienced by nurses.

ELIGIBILITY:
Inclusion Criteria:

* Employed as a registered nurse at Mayo Clinic Rochester or Mayo Clinic Florida.
* Primary work assignment is one of the following: medical-surgical units, operating and recovery rooms, emergency room, intensive/cardiac care units, or other special care units (including neonatal intensive care units and newborn nurseries).
* Proficient in written and spoken English.
* Able to provide written informed consent.

Exclusion Criteria:

- Any exception to above criteria.

Ages: 20 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Registered Nurses (RNs) at Mayo Clinic from Emergency Department, Intensive Care Units (including neonatal), selected Medical/Surgical units, and Inpatient Psychiatry. RNs from Inpatient Psychiatry will be recruited only from Mayo Rochester.
Sampling Method: Non-Probability Sample
Enrollment: 531 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Maslach Burnout Inventory-Human Services Survey (MBI-HSS) | Baseline, 3 months, 6 months, 9 months, 12 months
  Self-reported Maslach Burnout Inventory-Human Services Survey (MBI-HSS) assess clinician well-being in dimensions of burnout, engagement, and professional satisfaction. 22-item questionnaire ranking job-related feeling on 0 to 6 scale; 0 = never had this feeling, 6 = every day had this feeling

SECONDARY OUTCOMES:
Change in Quick Inventory of Depressive Symptomatology (QIDS-SR) | Baseline, 3 months, 6 months, 9 months, 12 months
  Self-reported Quick Inventory of Depressive Symptomatology (QIDS-SR) is a 16-item questionnaire that rates depression symptoms over the past seven days on an individual question scale of 0 to 3. Total scores range from 0 to 27 with higher scores indicating greater severity of depressive symptoms.
Change in LASA Quality of Life Scale | Baseline, 3 months, 6 months, 9 months, 12 months
  Linear Analogue Self-Assessment (LASA) 6-item questionnaire that assess feelings during the past week on an individual question scale of 0 to 10; 0 = as bad as it can be, 10 = as good as it can be. Total scores range 6-60 with higher scores indicating better perception of quality of life.
Sense of belonging | Baseline
  Measured using a 2- item self-reported questionnaire on sense of belonging to the nursing unit and hospital on an individual question scale of 0 to 4; 0=no opinion, 4=very strong. Total scores range from 0 to 8 with higher score indicating a greater sense of belonging.
Change in Food Intake Questionnaire | Baseline, 3 months, 6 months, 9 months, 12 months
  Measured using a self-reported multifactor food intake 16-item questionnaire that assess how many times per day, week or month subjects ate each food on a scale of never, 1-3 times last month, 1-2 times per week, 3-4 times per week, 5-6 times per week, 1 time per day, 2 times per day, 3 times per day, 4 or more times per day
Sleep quality | Every day over 12-month study period
  Measures by smartwatch that is worn daily by the subject reported in hours of sleep
Daily heart rate | 12 months
  Measured by smartwatch that is worn daily by the subject reported in beats per minute
Daily physical activity | 12 months
  Measured by smartwatch that is worn daily by the subject reported in time spent in activity (minutes)
Daily step count | 12 months
  Measured by smartwatch that is worn daily by the subject reported in number of steps per day

CONTACTS AND LOCATIONS:
Overall Officials: Arjun P. Athreya, Ph.D., M.S., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilton AR, Sheffield K, Wilkes Q, Chesak S, Pacyna J, Sharp R, Croarkin PE, Chauhan M, Dyrbye LN, Bobo WV, Athreya AP. The Burnout PRedictiOn Using Wearable aNd ArtIficial IntelligEnce (BROWNIE) study: a decentralized digital health protocol to predict burnout in registered nurses. BMC Nurs. 2024 Feb 13;23(1):114. doi: 10.1186/s12912-024-01711-8. PMID 38347557

DOCUMENTS (1):
  • Informed Consent Form (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT05481138/ICF_000.pdf